CLINICAL TRIAL: NCT00654173
Title: A 12-Week, Randomized, Open-Label, 3 Arm Parallel Group, Multicenter, Phase IIIb Study Comparing the Efficacy and Safety of Rosuvastatin With Atorvastatin and Simvastatin Achieving NCEP ATP III LDL-C Goals in High Risk Subjects With Hypercholesterolaemia in the Managed Care Setting.
Brief Title: Comparing the Efficacy and Safety of Rosuvastatin With Atorvastatin and Simvastatin (SOLAR)
Acronym: SOLAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Elisabeth Björk, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4522US/0003; D3560L00023
Record Dates: First submitted 2008-03-26; First posted 2008-04-07 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Hypercholesterolemia
Keywords: Cholesterol; low density lipoproteins; dyslipidaemia; Rosuvastatin; Crestor; Atorvastatin; Lipitor; Zocor; simvastatin
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias | interventions — Rosuvastatin Calcium; Simvastatin; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Rosuvastatin
  Interventions: Drug: Rosuvastatin
- 2 (Active Comparator): Simvastatin
  Interventions: Drug: Simvastatin
- 3 (Active Comparator): Atorvastatin
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Rosuvastatin
  Other Names: Crestor
  Arms: 1
Drug: Simvastatin
  Other Names: Zocor
  Arms: 2
Drug: Atorvastatin
  Other Names: Lipitor
  Arms: 3

SUMMARY:
The purpose of this study is to compare the efficacy and safety of rosuvastatin with simvastatin and atorvastatin in reducing levels of low density lipoprotein cholesterol in subjects with hypercholesterolaemia

ELIGIBILITY:
Inclusion Criteria:

* Member of managed care plan for hypercholesterolemia
* Fasting blood lipid levels as defined by the protocol
* Diagnosis of coronary heart disease, diabetes, or atherosclerotic disease, or presence of multiple risk factors giving high risk of coronary heart disease

Exclusion Criteria:

* The use of lipid lowering drugs or dietary supplements after Visit 1.
* Active arterial disease eg Unstable angina, or recent arterial surgery
* Blood lipid levels above the limits defined in the protocol.
* Uncontrolled hypertension, hypothyroidism, alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4444 (Actual)
Dates: Start 2002-06; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who achieve low density lipoprotein cholesterol goals while receiving treatment with rosuvastatin, compared to subjects receiving treatment with simvastatin or atorvastatin. | 6 weeks

SECONDARY OUTCOMES:
Percentage changes in other blood lipid levels while receiving treatment with rosuvastatin, compared to subjects receiving treatment with simvastatin or atorvastatin | 6 & 12 weeks
Safety: adverse events & abnormal laboratory markers | 6 & 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alex Gold, MD, Principal Investigator — AstraZeneca; Russell Esterline, Study Director — AstraZeneca